CLINICAL TRIAL: NCT03479242
Title: To Study Diabetic Foot Ulcer Recurrence With Trans Epidermal Water Loss Measured With Derma Lab
Brief Title: Diabetic Foot Ulcer Recurrence: Pilot Study
Acronym: DFUCO
Status: Terminated | Type: Observational
Why Stopped: Insufficient staffing
Sponsor: Indiana University (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Chandan Sen, Professor, Indiana University
Other Study IDs: 1808823394
Record Dates: First submitted 2018-01-25; First posted 2018-03-27 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Diabetic Foot; Ulcer Foot
MeSH Terms: conditions — Diabetic Foot; Foot Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no interventions — no interventions are planned

SUMMARY:
In this prospective pilot study, patients with DFU visiting the Indiana University Comprehensive Wound Center will be enrolled. Patients enrolled in the study will be followed for 16 weeks for wound closure(Phase A), and will then begin Phase B where TEWL measurements and wound recurrence will be followed up for up to 12 weeks.

DETAILED DESCRIPTION:
Diabetes impairs immune defenses such that the ability to fight wound infection is weakened. Thus, infection is a major problem in diabetic foot ulcers (DFUs) . Biofilms are estimated to account for 60% of chronic wound infections6. In biofilm bacteria are encased within extra polymeric substance (EPS) and become recalcitrant to antimicrobials and host defenses.In the biofilm form, bacteria may not form colony. Thus, standard clinical techniques like CFU to detect infection may not detect biofilm infection. Thus, biofilm infection may be viewed as a silent threat in wound care. Using a preclinical swine model of mixed species wound biofilm infection, we struck an unusual observation. Although biofilm infection may or may not influence the rate of wound closure as measured by standard planimetry, it inevitably compromises the functional property of the repaired skin. The wound may close as evaluated visually, but that closed wound lacks barrier function. Such pathology is caused by the perturbation of epithelial junctional proteins in response to biofilm infection. While detecting the biofilm directly is readily not possible at present in the wound clinics, compromised barrier function of the repaired skin can be detected at the point of care of the measurement of trans-epidermal water loss (TEWL). This pilot study, we propose, many DFUs that are currently served with a CLOSED clinical decision may have had a history of biofilm infection and therefore remained functionally open.

Considering that such incomplete wound closure may have a higher risk of wound recidivism, it becomes critically important that wound closure decisions be guided by functional tests in addition to factors currently considered. Importantly, substantial change in health impact may be achieved by a simple functional test as implemented by the measurement of trans epidermal water loss (TEWL). TEWL can be performed by clinical staff at the point of care within 15 minutes with minimum training using inexpensive hand- held pen like commercial gadgets approved for clinical use.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Willing to comply with protocol instructions, including all study visits and study activities.
3. Diabetic foot ulcers
4. Adequate arterial blood flow as evidenced by at least one of the following:

   1. TCOM > 30 mmHg
   2. Ankle-brachial index ≥0.7
   3. Toe pressure > 30 mmHg

Exclusion Criteria:

1. Individuals who are deemed unable to understand the procedures, risks and benefits of the study, (i.e. unable to provide informed consent)
2. Wounds closed or to be closed by flap or graft coverage
3. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 clinically diagnosed infected DFU patients will be recruited for this study in Phase A.Based on the expectation that 89% of these wounds will heal within 16 weeks of enrollment, 26 of these patients will continue with the study for Phase B.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Functional skin closure in DFU in relation to biofilm infection | 7 months
  TEWL will be measured to check for functional wound closure and see if DFU recidivism is high in subjects with a history of biofilm infection

CONTACTS AND LOCATIONS:
Overall Officials: Chandan K Sen, PhD, Principal Investigator — Professor
Locations (1):
- IU Health Methodist Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Roy S, Elgharably H, Sinha M, Ganesh K, Chaney S, Mann E, Miller C, Khanna S, Bergdall VK, Powell HM, Cook CH, Gordillo GM, Wozniak DJ, Sen CK. Mixed-species biofilm compromises wound healing by disrupting epidermal barrier function. J Pathol. 2014 Aug;233(4):331-343. doi: 10.1002/path.4360. Epub 2014 May 27. PMID 24771509
- See also: 1. Ahmed AS, Antonsen EL. Immune and vascular dysfunction in diabetic wound healing. J Wound Care. 2016;25 Suppl 7:S35-46 — https://www.ncbi.nlm.nih.gov/pubmed/29027849
- See also: 2. Aye M, Masson EA. Dermatological care of the diabetic foot. Am J Clin Dermatol. 2002;3:463-474 — https://www.ncbi.nlm.nih.gov/pubmed/?term=2.%09Aye+M%2C+Masson+EA.+Dermatological+care+of+the+diabetic+foot.+Am+J+Clin+Dermatol.+2002%3B3%3A463-474